CLINICAL TRIAL: NCT03193502
Title: Efficacy and Safety of Rivaroxaban in the Management of Acute Non-neoplastic Portal Vein Thrombosis in HCV Related Compensated Cirrhosis
Brief Title: Efficacy and Safety of Rivaroxaban in the Management of Acute Non-neoplastic PVT Compensated Cirrhosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amr Hanafy
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Portal Vein thrombosis (Experimental): rivaroxaban
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: rivaroxaban — rivaroxaban
  Other Names: xarelto

SUMMARY:
-Rivaroxaban is factor Xa inhibitor

DETAILED DESCRIPTION:
PVT is a common complication of liver cirrhosis

ELIGIBILITY:
Inclusion Criteria:

* Acute PVT

Exclusion Criteria:

* Malignant PVT
* Bleeding disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with recanalized portal vein | 6 months
  recanalization of portal vein

CONTACTS AND LOCATIONS:
Overall Officials: Amr Hanafy, Professor, Principal Investigator — Hepatology unit - Zagazig University; Mohamed Basha, Consultant, Study Director — Radiology Dept - Zagazig University; Sherief Abd-elsalam, consultant, Study Chair — Hepatology - Gastroenterology - Tanta University
Locations (1):
- Tropical medicine dept.-Tanta university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided